CLINICAL TRIAL: NCT04745013
Title: A Multi-center, Investigator-blinded, Randomized, 12-month, Parallel-group, Study to Compare the Clinical and Cost Efficacy of a New Hybrid Exercise Intervention PRIORITY Versus Usual Care
Brief Title: PeRsonalIzed remOtely Guided Preventive exeRcIse Therapy for a healThY Heart
Acronym: PRIORITY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Collaborators: Hasselt University (Other); University Hospital, Antwerp (Other); University Ghent (Other); Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Véronique Cornelissen, Professor, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: T004420N
Record Dates: First submitted 2021-02-04; First posted 2021-02-09 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Heart Failure With Preserved Ejection Fraction
MeSH Terms: interventions — Health Priorities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRIORITY (Experimental): Patients randomized to the hybrid exercise intervention (PRIORITY) will receive a personalized exercise prescription generated by the EXPERT tool which will then be person-tailored by the physiotherapist during one-on-one physical activity consultation. Over a period of one year, patients will participate in 18 supervised center-based exercise sessions in adjunct to a remotely monitored and guided home-based exercise intervention.
  Interventions: Behavioral: PRIORITY
- Usual care (Placebo Comparator): The usual care group will receive from the physiotherapist a personalized written exercise prescription that includes an individually tailored recommendation on frequency, intensity, type, time and volume of exercise. This exercise prescription will be generated by means of the EXPERT tool. No counselling or guidance on objective measures of physical activity by means of wearables or platform will be provided.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: PRIORITY — PeRsonalIzed remOtely guided preventive exeRcIse therapy for a healThY heart
  Arms: PRIORITY
Behavioral: Usual care — Only a written personalized exercise prescription will be provided.
  Arms: Usual care

SUMMARY:
In the PRIORITY study, we aim to provide the clinical evidence base for the use of a new hybrid exercise intervention, which includes remotely guided home-based exercise, as an accessible, clinical and cost-effective treatment to prevent the deleterious effects of sedentary aging on the heart and forestall the development and progression towards overt HFpEF.

ELIGIBILITY:
Inclusion Criteria: Men and women (HF stage A) aged > 30 yrs:

* treated or untreated patients with hypertension (blood pressure 130/80 - 159/99 mmHg) AND/OR
* Patients with prediabetes (impaired fasting glucose and/or insulin resistance) with either:

Fasting plasma glucose: 100 to 125 mg/dL (5.6-6.9 mmol/L) Hemoglobine A1c: 5.7% to 6.4% Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) index above 75% of population distribution (>2.0) AND/OR

* Patients with obesity with 30 kg/m² ≥ body mass index ≤ 42 kg/m²
* Patients with subclinical signs of diastolic dysfunction without symptoms (HF Stage B disease)
* Men and women with diagnosis of HF stage C: i.e. patients who have a total score ≥ 5 points according to the recent recommendation paper on how to diagnose heart failure with preserved ejection fraction from the Heart failure Association of ESC.

All participants should be on optimal medical treatment and stable with regard to symptoms and pharmacotherapy for at least 4 weeks before enrollment in the study. All participants should have internet access at home.

Exclusion Criteria:

* significant illness during the last 6 weeks
* known severe ventricular arrhythmia with functional or prognostic significance
* significant myocardial ischemia, hemodynamic deterioration or exercise-induced arrhythmia at baseline testing
* co-morbidity that may significantly negatively influence one-year prognosis
* functional or mental disability that may limit execution of prescribed exercise
* severe chronic obstructive pulmonary disease (FEV1 < 50%)
* NYHA class IV
* participation in another clinical interventional trial
* cognitive limitation

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes in cardiorespiratory fitness | 1- and 2-year follow-up
  Changes in cardiorespiratory fitness measured as pVO2 during a CPET until exhaustion

CONTACTS AND LOCATIONS:
Overall Officials: Véronique Cornelissen, PhD, Principal Investigator — KU Leuven
Locations (3):
- Belgium (3):
  - UZA, Antwerp
  - Jessa Hospital Hasselt, Hasselt
  - UHasselt, Hasselt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] De Wilde C, Bekhuis Y, Kuznetsova T, Claes J, Claessen G, Coninx K, Decorte E, De Smedt D, Hansen D, Lannoo M, Van Craenenbroeck EM, Verhaeghe N, Cornelissen VA. Personalized remotely guided preventive exercise therapy for a healthy heart (PRIORITY): protocol for an assessor-blinded, multicenter randomized controlled trial. Front Cardiovasc Med. 2023 Jun 29;10:1194693. doi: 10.3389/fcvm.2023.1194693. eCollection 2023. PMID 37456813